CLINICAL TRIAL: NCT02993757
Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Gardasil® in Healthy Subjects Aged 9 to 13 Years in Malaysia
Brief Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Gardasil®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CYD67; U1111-1161-3376 (Other: WHO); 2019-003135-36 (EudraCT Number)
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Human Papillomavirus Disease
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; Human Papillomavirus Disease; CYD Dengue Vaccine; Dengvaxia®; Gardasil®
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Dengue Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYD Dengue Vaccine + Gardasil (Concomitant Administration) (Experimental): Dengue immune participants received 3 doses of CYD dengue vaccine 0.5 milliliter (mL) subcutaneously (SC) at Day 0, Month 6, and Month 12; whereas dengue non-immune participants received only 2 doses of CYD vaccine at Day 0 and Month 6. Both immune and non-immune participants received 2 doses of Gardasil vaccine 0.5 mL Intramuscular (IM), concomitantly with the first 2 doses of CYD dengue vaccine.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Human Papillomavirus Quadrivalent [Types 6, 11, 16, and 18] Vaccine, Recombinant.
- CYD Dengue Vaccine + Gardasil (Sequential Administration) (Experimental): Dengue immune participants received 3 doses of CYD dengue vaccine 0.5 mL SC at Month 1, Month 7, and Month 13; whereas dengue non-immune participants received only 2 doses of CYD vaccine at Month 1 and Month 7. Both immune and non-immune participants received 2 doses of Gardasil vaccine 0.5 mL IM at Day 0 and Month 6 sequentially (i.e., one month before) to each of the first 2 doses of CYD dengue vaccine.
  Interventions: Biological: CYD Dengue Vaccine; Biological: Human Papillomavirus Quadrivalent [Types 6, 11, 16, and 18] Vaccine, Recombinant.

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 mL, SC injection at Day 0, Month 6 and 12, respectively.
  Other Names: Dengvaxia®
  Arms: CYD Dengue Vaccine + Gardasil (Concomitant Administration)
Biological: CYD Dengue Vaccine — 0.5 mL, SC injection at Month 1, 7 and 13, respectively.
  Other Names: Dengvaxia®
  Arms: CYD Dengue Vaccine + Gardasil (Sequential Administration)
Biological: Human Papillomavirus Quadrivalent [Types 6, 11, 16, and 18] Vaccine, Recombinant. — 0.5 mL, IM injection at Day 0 and Month 6, respectively.
  Other Names: Gardasil®

SUMMARY:
The aim of the study was to assess the safety and immunogenicity of the CYD dengue vaccine and Gardasil (Human Papillomavirus Quadrivalent [Types 6, 11, 16, and 18] Vaccine, Recombinant) when administered concomitantly or sequentially.

Primary objectives:

* To demonstrate that the humoral immune response (in terms of geometric mean titers [GMTs]) to Gardasil after concomitant administration was non-inferior to sequential administration with the CYD dengue vaccine measured 28 days after the last dose of Gardasil.
* To demonstrate that the humoral immune response to the CYD dengue vaccine after concomitant administration was non-inferior to sequential administration with Gardasil measured 28 days after the last dose of the CYD dengue vaccine.

Secondary Objectives:

* To demonstrate that the humoral immune response (in terms of seroconversion) to Gardasil vaccine after concomitant administration was non-inferior to sequential administration with the CYD dengue vaccine measured 28 days after the last dose of Gardasil.
* To describe the humoral immune response to Gardasil at baseline and after each dose of Gardasil in each and any group.
* To describe the humoral immune response to the CYD dengue vaccine at baseline and after each dose of the CYD dengue vaccine in each and any group.
* To describe the safety of Gardasil and the CYD dengue vaccine after each and any dose in each group.

DETAILED DESCRIPTION:
Participants received 3 doses of CYD dengue vaccine and 2 doses of Gardasil administered either concomitantly or sequentially.

The study activities were put on hold for several months (up to 6 months for some participants) to obtain the approval of Protocol Amendment 1 by the competent authorities and completed the associated logistic tasks. Due to this protocol amendment as per Independent Data Monitoring Committee recommendation, only previously dengue immune participants (seropositive for dengue before vaccination) were eligible to complete the vaccination schedule. Dengue non-immune participants (seronegative for dengue before vaccination) did not receive any additional CYD dengue vaccine injections, but were followed for safety up to 6 months after the last injection.

Due to the change in amendment 1, the number of evaluable dengue immune participants at baseline did not meet the predefined number of participants that would have allowed for a global power of at least 80% for non-inferiority testing of Gardasil vaccine and CYD dengue vaccine (121 per group for the co-primary objectives and 194 per group for the secondary objectives).

All participants were assessed for immunogenicity and safety. Safety assessments included solicited reactions within 7 or 14 days after each injection, unsolicited adverse events (AEs) within 28 days after each injection, non-serious AEs of Special Interests (AESIs) within 7 days after each injection, and serious adverse events including AESI and hospitalized virologically-confirmed dengue cases during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 9 to 13 years (i.e., from the day of the 9th birthday to the day prior to the 14th birthday) on the day of inclusion.
* Informed consent form (ICF) or Assent form (AF) had been signed and dated by the participant (based on local regulations), and/or ICF had been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* Participant (or participant and parent[s] or another legally acceptable representative) was (were) able to attend all scheduled visits and complied with all trial procedures.
* Participant in good health, based on medical history, and physical examination.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female had to be pre-menarche, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Previous vaccination against dengue disease with the trial vaccine.
* Previous vaccination against human papillomavirus (HPV) disease with either the trial vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency (including human immunodeficiency virus infection with impaired immune function); or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of HPV infection, confirmed either clinically, serologically, or microbiologically as reported by participant or parent(s) or another legally acceptable representative.
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Thrombocytopenia, contraindicating IM vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction that, based on investigator's judgment, might interfered with the participant's ability to comply with trial procedures.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfered with trial conduct or completion.
* Identified as an Investigator or employee of the Investigator with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Self-reported Hepatitis B, Hepatitis C infection.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 528 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (5):
- Malaysia (5):
  - Sanofi Pasteur Investigational Site 004, Klang
  - Sanofi Pasteur Investigational Site 005, Kuala Lumpur
  - Sanofi Pasteur Investigational Site 001, Kuala Lumpur
  - Sanofi Pasteur Investigational Site 003, Kuantan
  - Sanofi Pasteur Investigational Site 002, Sibu

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Hassan J, Toh TH, Sivapunniam SK, Hasim R, Ghazali NF, Sulaiman S, Koh MT, Meyer S, Toh ML, Zocchetti C, Vigne C, Mascarenas C. Immunogenicity and Safety of a Tetravalent Dengue Vaccine Administered Concomitantly or Sequentially With Quadrivalent Human Papillomavirus Vaccine in Boys and Girls 9-13 Years of Age in Malaysia: A Phase IIIb, Randomized, Open-label Study. Pediatr Infect Dis J. 2021 Aug 1;40(8):774-781. doi: 10.1097/INF.0000000000003164. PMID 34250977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 01 December 2016 to 16 April 2017 at 5 centers in Malaysia. A total of 528 participants were enrolled and randomized in study.
Pre-assignment Details: As per protocol amendment 1, only dengue immune participants at baseline completed the dengue vaccination schedule and received 3 doses of CYD dengue vaccine, whereas the dengue non-immune participants received only 2 doses of CYD dengue vaccine. All participants were followed for safety up to 6 months after the last vaccination.
Groups:
- CYD Dengue Vaccine + Gardasil (Concomitant Administration): Dengue immune participants (i.e., titers greater than or equal to (>=)10 (1/dilution [dil]) for at least one serotype with the parental dengue virus strains in the baseline sample) received 3 doses of CYD dengue vaccine 0.5 milliliter (mL) subcutaneously (SC) at Day 0, Month 6, and Month 12; whereas dengue non-immune participants (i.e., titers less than (<)10 (1/dil) for all serotypes with parental dengue virus strains with available and "valid" results in the baseline sample) received only 2 doses of CYD vaccine at Day 0 and Month 6. Both immune and non-immune participants received 2 doses of Gardasil vaccine 0.5 mL Intramuscular (IM), concomitantly with the first 2 doses of CYD dengue vaccine.
- CYD Dengue Vaccine + Gardasil (Sequential Administration): Dengue immune participants (i.e., titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains in the baseline sample) received 3 doses of CYD dengue vaccine 0.5 mL SC at Month 1, Month 7, and Month 13; whereas dengue non-immune participants (i.e., titers <10 (1/dil) for all serotypes with parental dengue virus strains with available and "valid" results in the baseline sample) received only 2 doses of CYD vaccine at Month 1 and Month 7. Both immune and non-immune participants received 2 doses of Gardasil vaccine 0.5 mL IM at Day 0 and Month 6 sequentially (i.e., one month before) to each of the first 2 doses of CYD dengue vaccine.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Started | 266 | 262
Safety Analysis Set (SafAS) (SafAS was defined as participants who had received at least 1 dose of study vaccines.) | 263 | 260
Completed | 102 | 84
Not Completed | 164 | 178
Not completed — Non compliance with the protocol | 155 | 170
Not completed — Lost to Follow-up | 1 | 0
Not completed — Voluntary withdraw not due adverse event | 8 | 8

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- CYD Dengue Vaccine + Gardasil (Concomitant Administration): Dengue immune participants received 3 doses of CYD dengue vaccine 0.5 mL SC at Day 0, Month 6, and Month 12; whereas dengue non-immune participants received only 2 doses of CYD vaccine at Day 0 and Month 6. Both immune and non-immune participants received 2 doses of Gardasil vaccine 0.5 mL IM, concomitantly with the first 2 doses of CYD dengue vaccine.
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration) | Total
Number analyzed (Participants) | 266 | 262 | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (1.20) | 10.5 (1.18) | 10.4 (1.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 172 | 347
  Male | 91 | 90 | 181
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Dengue Seropositivity Status [Count of Participants; unit: Participants] — Dengue immune participants were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains in the baseline sample.
  Dengue non-immune participants were defined as participants with titers <10 (1/dil) for all serotypes with parental dengue virus strains with available and "valid" results in the baseline sample.
  Participants
    Dengue immune | 109 | 88 | 197
    Dengue non-immune | 157 | 174 | 331

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) Against Each Gardasil Vaccine Human Papillomavirus (HPV) Antigen (HPV-6, HPV-11, HPV-16, HPV-18) 28 Days After Last Gardasil Vaccination in the Previously Dengue Immune Participants
Description: GMTs (measured in milli-Merck Units per mL [mMU/mL]) against each Gardasil HPV antigen (HPV-6, HPV-11, HPV-16, HPV-18) were assessed using competitive Luminex immunoassay (cLIA) method. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains.
Time Frame: 28 days after the last Gardasil vaccination
Population: Analysis was performed on full analysis set (FAS) that included subset of participants who received at least one dose of each of study vaccines (CYD and Gardasil), analyzed by baseline dengue status & vaccine group randomized. Here,'overall number of participants analyzed' = participants evaluable and had available data for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 104 | 86
mMU/mL
  HPV-6 | 420 [327 to 539] | 428 [314 to 583]
  HPV-11 | 1288 [1089 to 1522] | 1601 [1323 to 1937]
  HPV-16 | 6221 [5093 to 7598] | 7629 [6142 to 9475]
  HPV-18 | 829 [682 to 1007] | 1042 [858 to 1266]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Antigen HPV-6; Test type: Other; GMT ratio = 0.982, 95% CI 2-sided [0.664 to 1.45]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Antigen HPV-11; Test type: Other; GMT ratio = 0.804, 95% CI 2-sided [0.626 to 1.03]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Antigen HPV-16; Test type: Other; GMT ratio = 0.815, 95% CI 2-sided [0.608 to 1.09]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Antigen HPV-18; Test type: Other; GMT ratio = 0.795, 95% CI 2-sided [0.603 to 1.05]

2. Primary Outcome: Geometric Mean Titers Against Each Parental Dengue Virus Serotype 28 Days After Third CYD Dengue Vaccination in the Previously Dengue Immune Participants
Description: The GMTs against each of the four parental dengue virus serotypes (1, 2, 3, and 4) of CYD dengue vaccine was assessed using the 50% plaque reduction neutralization test (PRNT50) assay. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains.
Time Frame: 28 days after third CYD dengue vaccination
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants evaluable and had available data for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer (1/dilution)
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 102 | 84
titer (1/dilution)
  Serotype 1 | 447 [303 to 659] | 453 [313 to 656]
  Serotype 2 | 561 [408 to 771] | 717 [526 to 977]
  Serotype 3 | 460 [354 to 596] | 549 [411 to 734]
  Serotype 4 | 323 [263 to 398] | 303 [255 to 359]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Serotype 1; Test type: Other; GMT ratio = 0.987, 95% CI 2-sided [0.574 to 1.70]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Serotype 2; Test type: Other; GMT ratio = 0.783, 95% CI 2-sided [0.500 to 1.22]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Serotype 3; Test type: Other; GMT ratio = 0.836, 95% CI 2-sided [0.568 to 1.23]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine + Gardasil (Concomitant Administration) vs CYD Dengue Vaccine + Gardasil (Sequential Administration); Serotype 4; Test type: Other; GMT ratio = 1.07, 95% CI 2-sided [0.813 to 1.40]

3. Secondary Outcome: Percentage of Participants With Seroconversion Against Each Gardasil HPV Antigen (HPV-6, HPV-11, HPV-16, HPV-18) 28 Days After Last Dose of Gardasil in the Previously Dengue Immune Participants
Description: Neutralizing antibodies against each Gardasil HPV antigen (HPV-6, HPV-11, HPV-16, HPV-18) was assessed using cLIA method. Seroconversion was defined as changing serostatus from seronegative at baseline to seropositive (participants with a pre-vaccination titer < lower limit of quantification [LLOQ] (mMU/mL) to a post-vaccination titer >=LLOQ) or >=4-fold rise in antibody titer if seropositive at baseline. The LLOQ for HPV-6 and HPV-16 was 11 mMU/mL, 8 mMU/mL for HPV-11, and 10 mMU/mL for HPV-18. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains.
Time Frame: 28 days after the last Gardasil vaccination
Population: Analysis was performed on FAS. Here, 'overall number of participants analyzed' = participants evaluable and had available data for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 103 | 81
percentage of participants
  HPV-6 | 98.1 [93.2 to 99.8] | 100.0 [95.5 to 100.0]
  HPV-11 | 100.0 [96.5 to 100.0] | 100.0 [95.5 to 100.0]
  HPV-16 | 100.0 [96.5 to 100.0] | 100.0 [95.5 to 100.0]
  HPV-18 | 100.0 [96.5 to 100.0] | 100.0 [95.5 to 100.0]

4. Secondary Outcome: Geometric Mean Titers Against Each Gardasil HPV Antigen (HPV-6, HPV-11, HPV-16, HPV-18) at Day 0 and 28 Days After Each Dose of Gardasil in the Previously Dengue Immune Participants
Description: The GMTs (measured in mMU/mL) against each Gardasil HPV antigen (HPV-6, HPV-11, HPV-16, HPV-18) was assessed using cLIA method. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains.
Time Frame: Day 0 (pre-vaccination) and 28 days after Gardasil vaccination 1 and 2
Population: Analysis was performed on FAS. Here, 'overall number of participants analyzed' = participants evaluable and had available data for this outcome measure and 'Number analyzed' = participants with available data for each specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 109 | 88
mMU/mL
  HPV-6: Day 0: number analyzed (Participants) | 108 | 82
  HPV-6: Day 0 | 5.70 [5.46 to 5.95] | 5.61 [5.46 to 5.77]
  HPV-6: 28 days post vaccination 1: number analyzed (Participants) | 107 | 88
  HPV-6: 28 days post vaccination 1 | 54.9 [45.0 to 66.9] | 61.8 [49.7 to 76.9]
  HPV-6: 28 days post vaccination 2: number analyzed (Participants) | 104 | 86
  HPV-6: 28 days post vaccination 2 | 420 [327 to 539] | 428 [314 to 583]
  HPV-11: Day 0: number analyzed (Participants) | 108 | 82
  HPV-11: Day 0 | 4.16 [3.92 to 4.41] | 4.00 [NA to NA] — The 95% confidence interval was not computable, since all participants had the same value.
  HPV-11: 28 days post vaccination 1: number analyzed (Participants) | 107 | 88
  HPV-11: 28 days post vaccination 1 | 58.1 [47.6 to 71.0] | 78.5 [62.5 to 98.6]
  HPV-11: 28 days post vaccination 2: number analyzed (Participants) | 104 | 86
  HPV-11: 28 days post vaccination 2 | 1288 [1089 to 1522] | 1601 [1323 to 1937]
  HPV-16: Day 0: number analyzed (Participants) | 108 | 82
  HPV-16: Day 0 | 5.62 [5.38 to 5.87] | 5.50 [NA to NA] — The 95% confidence interval was not computable, since all participants had the same value.
  HPV-16: 28 days post vaccination 1: number analyzed (Participants) | 107 | 88
  HPV-16: 28 days post vaccination 1 | 148 [119 to 185] | 150 [116 to 193]
  HPV-16: 28 days post vaccination 2: number analyzed (Participants) | 104 | 86
  HPV-16: 28 days post vaccination 2 | 6221 [5093 to 7598] | 7629 [6142 to 9475]
  HPV-18: Day 0: number analyzed (Participants) | 108 | 82
  HPV-18: Day 0 | 5.26 [5.03 to 5.50] | 5.06 [4.94 to 5.18]
  HPV-18: 28 days post vaccination 1: number analyzed (Participants) | 107 | 88
  HPV-18: 28 days post vaccination 1 | 23.5 [18.7 to 29.4] | 31.6 [24.9 to 40.0]
  HPV-18: 28 days post vaccination 2: number analyzed (Participants) | 104 | 86
  HPV-18: 28 days post vaccination 2 | 829 [682 to 1007] | 1042 [858 to 1266]

5. Secondary Outcome: Geometric Mean Titers Against Each Dengue Virus Serotype of CYD Dengue Vaccine at Day 0 and 28 Days After Each Dose of CYD Dengue Vaccination in the Previously Dengue Immune Participants
Description: The GMTs against each of the four parental dengue virus serotypes (1, 2, 3, and 4) of CYD dengue vaccine was assessed using the PRNT50 assay. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains.
Time Frame: Day 0 (pre-vaccination) and 28 days after each CYD dengue vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: titer (1/dilution)
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 109 | 88
titer (1/dilution)
  Serotype 1: Day 0 | 62.3 [40.7 to 95.5] | 81.5 [49.4 to 135]
  Serotype 1: 28 days post vaccination 1: number analyzed (Participants) | 107 | 88
  Serotype 1: 28 days post vaccination 1 | 382 [245 to 597] | 449 [268 to 752]
  Serotype 1: 28 days post vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 1: 28 days post vaccination 2 | 403 [270 to 602] | 529 [342 to 819]
  Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 1: 28 days post vaccination 3 | 447 [303 to 659] | 453 [313 to 656]
  Serotype 2: Day 0 | 110 [75.5 to 160] | 130 [84.0 to 201]
  Serotype 2: 28 days post-vaccination 1: number analyzed (Participants) | 107 | 88
  Serotype 2: 28 days post-vaccination 1 | 750 [500 to 1124] | 848 [541 to 1330]
  Serotype 2: 28 days post-vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 2: 28 days post-vaccination 2 | 728 [519 to 1019] | 937 [654 to 1342]
  Serotype 2: 28 days post-vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 2: 28 days post-vaccination 3 | 561 [408 to 771] | 717 [526 to 977]
  Serotype 3: Day 0: number analyzed (Participants) | 109 | 87
  Serotype 3: Day 0 | 72.3 [52.7 to 99.2] | 96.7 [64.9 to 144]
  Serotype 3: 28 days post-vaccination 1: number analyzed (Participants) | 106 | 88
  Serotype 3: 28 days post-vaccination 1 | 432 [304 to 614] | 517 [355 to 755]
  Serotype 3: 28 days post-vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 3: 28 days post-vaccination 2 | 389 [299 to 506] | 543 [403 to 731]
  Serotype 3: 28 days post-vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 3: 28 days post-vaccination 3 | 460 [354 to 596] | 549 [411 to 734]
  Serotype 4: Day 0 | 26.3 [18.8 to 36.7] | 23.7 [16.2 to 34.8]
  Serotype 4: 28 days post-vaccination 1: number analyzed (Participants) | 107 | 88
  Serotype 4: 28 days post-vaccination 1 | 330 [234 to 464] | 286 [204 to 401]
  Serotype 4: 28 days post-vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 4: 28 days post-vaccination 2 | 284 [229 to 352] | 282 [225 to 353]
  Serotype 4: 28 days post-vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 4: 28 days post-vaccination 3 | 323 [263 to 398] | 303 [255 to 359]

6. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers Against Each of the 4 Dengue Virus Serotypes of CYD Dengue Vaccine at Day 0 And 28 Days After Each Dose of CYD Dengue Vaccination in the Previously Dengue Immune Participants
Description: Dengue neutralizing antibody levels against each of the 4 dengue virus serotypes (1, 2, 3, and 4) was measured by PRNT50. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains.
Time Frame: Day 0 (pre-vaccination) and 28 days after each CYD dengue vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 109 | 88
percentage of participants
  Serotype 1: Day 0 | 66.1 [56.4 to 74.9] | 72.7 [62.2 to 81.7]
  Serotype 1: 28 days post vaccination 1: number analyzed (Participants) | 107 | 88
  Serotype 1: 28 days post vaccination 1 | 91.6 [84.6 to 96.1] | 90.9 [82.9 to 96.0]
  Serotype 1: 28 days post vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 1: 28 days post vaccination 2 | 96.2 [90.4 to 98.9] | 95.4 [88.6 to 98.7]
  Serotype 1: 28 days post vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 1: 28 days post vaccination 3 | 95.1 [88.9 to 98.4] | 100.0 [95.7 to 100.0]
  Serotype 2: Day 0 | 83.5 [75.2 to 89.9] | 81.8 [72.2 to 89.2]
  Serotype 2: 28 days post-vaccination 1: number analyzed (Participants) | 107 | 88
  Serotype 2: 28 days post-vaccination 1 | 93.5 [87.0 to 97.3] | 92.0 [84.3 to 96.7]
  Serotype 2: 28 days post-vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 2: 28 days post-vaccination 2 | 99.0 [94.8 to 100.0] | 97.7 [91.9 to 99.7]
  Serotype 2: 28 days post-vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 2: 28 days post-vaccination 3 | 97.1 [91.6 to 99.4] | 98.8 [93.5 to 100.0]
  Serotype 3: Day 0: number analyzed (Participants) | 109 | 87
  Serotype 3: Day 0 | 89.0 [81.6 to 94.2] | 86.2 [77.1 to 92.7]
  Serotype 3: 28 days post-vaccination 1: number analyzed (Participants) | 106 | 88
  Serotype 3: 28 days post-vaccination 1 | 96.2 [90.6 to 99.0] | 97.7 [92.0 to 99.7]
  Serotype 3: 28 days post-vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 3: 28 days post-vaccination 2 | 100.0 [96.5 to 100.0] | 100.0 [95.8 to 100.0]
  Serotype 3: 28 days post-vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 3: 28 days post-vaccination 3 | 99.0 [94.7 to 100.0] | 100.0 [95.7 to 100.0]
  Serotype 4: Day 0 | 59.6 [49.8 to 68.9] | 54.5 [43.6 to 65.2]
  Serotype 4: 28 days post-vaccination 1: number analyzed (Participants) | 107 | 88
  Serotype 4: 28 days post-vaccination 1 | 93.5 [87.0 to 97.3] | 98.9 [93.8 to 100.0]
  Serotype 4: 28 days post-vaccination 2: number analyzed (Participants) | 104 | 87
  Serotype 4: 28 days post-vaccination 2 | 100.0 [96.5 to 100.0] | 100.0 [95.8 to 100.0]
  Serotype 4: 28 days post-vaccination 3: number analyzed (Participants) | 102 | 84
  Serotype 4: 28 days post-vaccination 3 | 100.0 [96.4 to 100.0] | 100.0 [95.7 to 100.0]

7. Secondary Outcome: Percentage of Participants With Neutralizing Antibody Titers Above Pre-defined Thresholds Against at Least 1,2,3,or4 Serotypes of CYD Dengue Vaccine at Day 0 And 28 Days After Each Dose of CYD Dengue Vaccination in Previously Dengue Immune Participants
Description: Dengue neutralizing antibody levels against each of the 4 dengue virus serotypes (1, 2, 3, and 4) was measured by PRNT50. Dengue immune participants at Baseline were defined as participants with titers >=10 (1/dil) for at least one serotype with the parental dengue virus strains. Percentage of participants with neutralizing antibody titers above pre-defined thresholds (>=10 and >=100 [1/dil]) against at least 1, 2, 3, or 4 serotypes of CYD dengue vaccine were reported.
Time Frame: Day 0 (pre-vaccination) and 28 days after each CYD dengue vaccination
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 109 | 88
percentage of participants
  At least 1 Serotype: Day 0: >=10 (1/dil) | 100.0 [96.7 to 100.0] | 100.0 [95.9 to 100.0]
  At least 1 Serotype: Day 0: >=100 (1/dil) | 90.8 [83.8 to 95.5] | 88.6 [80.1 to 94.4]
  At least 1 Serotype:post vaccination 1:>=10(1/dil): number analyzed (Participants) | 107 | 88
  At least 1 Serotype:post vaccination 1:>=10(1/dil) | 97.2 [92.0 to 99.4] | 100.0 [95.9 to 100.0]
  At least 1 Serotype:post vaccination1:>=100(1/dil): number analyzed (Participants) | 107 | 88
  At least 1 Serotype:post vaccination1:>=100(1/dil) | 95.3 [89.4 to 98.5] | 96.6 [90.4 to 99.3]
  At least 1 Serotype:post vaccination 2:>=10(1/dil): number analyzed (Participants) | 104 | 87
  At least 1 Serotype:post vaccination 2:>=10(1/dil) | 100.0 [96.5 to 100.0] | 100.0 [95.8 to 100.0]
  At least 1 Serotype:post vaccination2:>=100(1/dil): number analyzed (Participants) | 104 | 87
  At least 1 Serotype:post vaccination2:>=100(1/dil) | 96.2 [90.4 to 98.9] | 98.9 [93.8 to 100.0]
  At least 1 Serotype:post vaccination 3:>=10(1/dil): number analyzed (Participants) | 102 | 84
  At least 1 Serotype:post vaccination 3:>=10(1/dil) | 100.0 [96.4 to 100.0] | 100.0 [95.7 to 100.0]
  At least 1 Serotype:post vaccination3:>=100(1/dil): number analyzed (Participants) | 102 | 84
  At least 1 Serotype:post vaccination3:>=100(1/dil) | 98.0 [93.1 to 99.8] | 97.6 [91.7 to 99.7]
  At least 2 Serotypes: Day 0: >=10 (1/dil) | 84.4 [76.2 to 90.6] | 81.8 [72.2 to 89.2]
  At least 2 Serotypes: Day 0: >=100 (1/dil) | 34.9 [26.0 to 44.6] | 39.8 [29.5 to 50.8]
  At least 2 Serotypes:post vaccination1:>=10(1/dil): number analyzed (Participants) | 107 | 88
  At least 2 Serotypes:post vaccination1:>=10(1/dil) | 94.4 [88.2 to 97.9] | 97.7 [92.0 to 99.7]
  At least 2Serotypes:post vaccination1:>=100(1/dil): number analyzed (Participants) | 107 | 88
  At least 2Serotypes:post vaccination1:>=100(1/dil) | 85.0 [76.9 to 91.2] | 80.7 [70.9 to 88.3]
  At least 2 Serotypes:post vaccination2:>=10(1/dil): number analyzed (Participants) | 104 | 87
  At least 2 Serotypes:post vaccination2:>=10(1/dil) | 100.0 [96.5 to 100.0] | 100.0 [95.8 to 100.0]
  At least 2Serotypes:post vaccination2:>=100(1/dil): number analyzed (Participants) | 104 | 87
  At least 2Serotypes:post vaccination2:>=100(1/dil) | 84.6 [76.2 to 90.9] | 92.0 [84.1 to 96.7]
  At least 2 Serotypes:post vaccination3:>=10(1/dil): number analyzed (Participants) | 102 | 84
  At least 2 Serotypes:post vaccination3:>=10(1/dil) | 100.0 [96.4 to 100.0] | 100.0 [95.7 to 100.0]
  At least 2Serotypes:post vaccination3:>=100(1/dil): number analyzed (Participants) | 102 | 84
  At least 2Serotypes:post vaccination3:>=100(1/dil) | 93.1 [86.4 to 97.2] | 94.0 [86.7 to 98.0]
  At least 3 Serotypes:Day 0: >=10 (1/dil) | 71.6 [62.1 to 79.8] | 69.3 [58.6 to 78.7]
  At least 3 Serotypes:Day 0: >=100 (1/dil) | 23.9 [16.2 to 33.0] | 27.3 [18.3 to 37.8]
  At least 3 Serotypes:post vaccination1:>=10(1/dil): number analyzed (Participants) | 107 | 88
  At least 3 Serotypes:post vaccination1:>=10(1/dil) | 92.5 [85.8 to 96.7] | 92.0 [84.3 to 96.7]
  At least 3Serotypes:post vaccination1:>=100(1/dil): number analyzed (Participants) | 107 | 88
  At least 3Serotypes:post vaccination1:>=100(1/dil) | 75.7 [66.5 to 83.5] | 73.9 [63.4 to 82.7]
  At least 3 Serotypes:post vaccination2:>=10(1/dil): number analyzed (Participants) | 104 | 87
  At least 3 Serotypes:post vaccination2:>=10(1/dil) | 99.0 [94.8 to 100.0] | 98.9 [93.8 to 100.0]
  At least 3Serotypes:post vaccination2:>=100(1/dil): number analyzed (Participants) | 104 | 87
  At least 3Serotypes:post vaccination2:>=100(1/dil) | 77.9 [68.7 to 85.4] | 86.2 [77.1 to 92.7]
  At least 3 Serotypes:post vaccination3:>=10(1/dil): number analyzed (Participants) | 102 | 84
  At least 3 Serotypes:post vaccination3:>=10(1/dil) | 97.1 [91.6 to 99.4] | 100.0 [95.7 to 100.0]
  At least 3Serotypes:post vaccination3:>=100(1/dil): number analyzed (Participants) | 102 | 84
  At least 3Serotypes:post vaccination3:>=100(1/dil) | 83.3 [74.7 to 90.0] | 88.1 [79.2 to 94.1]
  At least 4 Serotypes:Day 0: >=10 (1/dil): number analyzed (Participants) | 109 | 87
  At least 4 Serotypes:Day 0: >=10 (1/dil) | 42.2 [32.8 to 52.0] | 43.7 [33.1 to 54.7]
  At least 4 Serotypes:Day 0: >=100 (1/dil): number analyzed (Participants) | 109 | 87
  At least 4 Serotypes:Day 0: >=100 (1/dil) | 6.4 [2.6 to 12.8] | 12.6 [6.5 to 21.5]
  At least 4 Serotypes:post vaccination1:>=10(1/dil): number analyzed (Participants) | 106 | 88
  At least 4 Serotypes:post vaccination1:>=10(1/dil) | 90.6 [83.3 to 95.4] | 89.8 [81.5 to 95.2]
  At least 4Serotypes:post vaccination1:>=100(1/dil): number analyzed (Participants) | 106 | 88
  At least 4Serotypes:post vaccination1:>=100(1/dil) | 60.4 [50.4 to 69.7] | 62.5 [51.5 to 72.6]
  At least 4 Serotypes:post vaccination2:>=10(1/dil): number analyzed (Participants) | 104 | 87
  At least 4 Serotypes:post vaccination2:>=10(1/dil) | 96.2 [90.4 to 98.9] | 94.3 [87.1 to 98.1]
  At least 4Serotypes:post vaccination2:>=100(1/dil): number analyzed (Participants) | 104 | 87
  At least 4Serotypes:post vaccination2:>=100(1/dil) | 67.3 [57.4 to 76.2] | 75.9 [65.5 to 84.4]
  At least 4 Serotypes:post vaccination3:>=10(1/dil): number analyzed (Participants) | 102 | 84
  At least 4 Serotypes:post vaccination3:>=10(1/dil) | 94.1 [87.6 to 97.8] | 98.8 [93.5 to 100.0]
  At least 4Serotypes:post vaccination3:>=100(1/dil): number analyzed (Participants) | 102 | 84
  At least 4Serotypes:post vaccination3:>=100(1/dil) | 72.5 [62.8 to 80.9] | 77.4 [67.0 to 85.8]

8. Secondary Outcome: Number of Participants Reporting Immediate Adverse Events (AEs) Following Vaccination With Gardasil or CYD Dengue Vaccine
Description: Any unsolicited systemic AE occurred during the first 30 minutes post-vaccination was recorded on the case report form (CRF) as immediate AE. At Visit 1 and Visit 4, participants from Group 1 received both Gardasil and CYD vaccination and participants from Group 2 received only Gardasil vaccination. At Visit 2 and Visit 5, only participants from Group 2 received CYD vaccination whereas the participants from Group 1 received no vaccination.
Time Frame: Within 30 minutes after any and each vaccination
Population: Analysis was performed on safety analysis set (SafAS) which included participants who have received at least one dose of the study vaccines. Here, 'Number analyzed' = participants with available data for each specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 263 | 260
Participants
  Post any vaccination | 0 | 3
  Post vaccination 1 (Visit 1) | 0 | 1
  Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 256
  Post CYD vaccination 1 (Visit 2) |  | 1
  Post vaccination 2 (Visit 4): number analyzed (Participants) | 257 | 256
  Post vaccination 2 (Visit 4) | 0 | 0
  Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Post CYD vaccination 2 (Visit 5) |  | 1
  Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Post CYD vaccination 3 (Visit 7) | 0 | 0

9. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions Following Vaccination With Gardasil or CYD Dengue Vaccine
Description: A solicited reaction (SR) was an adverse reaction (AR) observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the CRF and considered as related to vaccination. Solicited injection site reactions included pain, erythema, and swelling.
Time Frame: Up to 7 days after any and each vaccination
Population: Analysis was performed on SafAS. Here, 'Number analyzed' = participants with available data for each specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 263 | 260
Participants
  Pain: Post any CYD/Gardasil vaccine: number analyzed (Participants) | 260 | 258
  Pain: Post any CYD/Gardasil vaccine | 206 | 193
  Pain: Post CYD/Gardasil vaccination 1: number analyzed (Participants) | 260 | 258
  Pain: Post CYD/Gardasil vaccination 1 | 163 | 157
  Pain: Post CYD/Gardasil vaccination 2: number analyzed (Participants) | 256 | 254
  Pain: Post CYD/Gardasil vaccination 2 | 151 | 141
  Pain: Post CYD vaccination 3: number analyzed (Participants) | 103 | 83
  Pain: Post CYD vaccination 3 | 33 | 24
  Erythema: Post any CYD/Gardasil vaccine: number analyzed (Participants) | 260 | 258
  Erythema: Post any CYD/Gardasil vaccine | 45 | 38
  Erythema: Post CYD/Gardasil vaccination 1: number analyzed (Participants) | 260 | 258
  Erythema: Post CYD/Gardasil vaccination 1 | 30 | 29
  Erythema: Post CYD/Gardasil vaccination 2: number analyzed (Participants) | 256 | 254
  Erythema: Post CYD/Gardasil vaccination 2 | 25 | 19
  Erythema: Post CYD vaccination 3: number analyzed (Participants) | 103 | 83
  Erythema: Post CYD vaccination 3 | 9 | 2
  Swelling: Post any CYD/Gardasil vaccine: number analyzed (Participants) | 260 | 258
  Swelling: Post any CYD/Gardasil vaccine | 43 | 31
  Swelling: Post CYD/Gardasil vaccination 1: number analyzed (Participants) | 260 | 258
  Swelling: Post CYD/Gardasil vaccination 1 | 22 | 22
  Swelling: Post CYD/Gardasil vaccination 2: number analyzed (Participants) | 256 | 254
  Swelling: Post CYD/Gardasil vaccination 2 | 30 | 18
  Swelling: Post CYD vaccination 3: number analyzed (Participants) | 103 | 83
  Swelling: Post CYD vaccination 3 | 9 | 3

10. Secondary Outcome: Number of Participants Reporting Solicited Systemic Reactions Following Vaccination With Gardasil or CYD Dengue Vaccine
Description: A SR was an AR observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the CRF and considered as related to vaccination. Solicited systemic reactions included fever, headache, malaise, myalgia, and asthenia. At Visit 1 and Visit 4, participants from Group 1 received both Gardasil and CYD vaccination and participants from Group 2 received only Gardasil vaccination. At Visit 2 and Visit 5, only participants from Group 2 received CYD vaccination whereas the participants from Group 1 received no vaccination.
Time Frame: Up to 14 days after any and each vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 263 | 260
Participants
  Fever: Post any vaccination: number analyzed (Participants) | 259 | 258
  Fever: Post any vaccination | 36 | 47
  Fever: Post vaccination 1 (Visit 1): number analyzed (Participants) | 257 | 258
  Fever: Post vaccination 1 (Visit 1) | 21 | 8
  Fever: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 255
  Fever: Post CYD vaccination 1 (Visit 2) |  | 15
  Fever: Post vaccination 2 (Visit 4): number analyzed (Participants) | 252 | 253
  Fever: Post vaccination 2 (Visit 4) | 10 | 11
  Fever: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Fever: Post CYD vaccination 2 (Visit 5) |  | 12
  Fever: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Fever: Post CYD vaccination 3 (Visit 7) | 8 | 6
  Headache: Post any vaccination: number analyzed (Participants) | 260 | 258
  Headache: Post any vaccination | 125 | 146
  Headache: Post vaccination 1 (Visit 1): number analyzed (Participants) | 260 | 258
  Headache: Post vaccination 1 (Visit 1) | 99 | 93
  Headache: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 255
  Headache: Post CYD vaccination 1 (Visit 2) |  | 73
  Headache: Post vaccination 2 (Visit 4): number analyzed (Participants) | 256 | 254
  Headache: Post vaccination 2 (Visit 4) | 61 | 70
  Headache: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Headache: Post CYD vaccination 2 (Visit 5) |  | 51
  Headache: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Headache: Post CYD vaccination 3 (Visit 7) | 15 | 17
  Malaise: Post any vaccination: number analyzed (Participants) | 260 | 258
  Malaise: Post any vaccination | 111 | 137
  Malaise: Post vaccination 1 (Visit 1): number analyzed (Participants) | 260 | 258
  Malaise: Post vaccination 1 (Visit 1) | 82 | 78
  Malaise: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 255
  Malaise: Post CYD vaccination 1 (Visit 2) |  | 69
  Malaise: Post vaccination 2 (Visit 4): number analyzed (Participants) | 256 | 254
  Malaise: Post vaccination 2 (Visit 4) | 57 | 54
  Malaise: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Malaise: Post CYD vaccination 2 (Visit 5) |  | 40
  Malaise: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Malaise: Post CYD vaccination 3 (Visit 7) | 20 | 17
  Myalgia: Post any vaccination: number analyzed (Participants) | 260 | 258
  Myalgia: Post any vaccination | 127 | 156
  Myalgia: Post vaccination 1 (Visit 1): number analyzed (Participants) | 260 | 258
  Myalgia: Post vaccination 1 (Visit 1) | 93 | 94
  Myalgia: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 255
  Myalgia: Post CYD vaccination 1 (Visit 2) |  | 63
  Myalgia: Post vaccination 2 (Visit 4): number analyzed (Participants) | 256 | 254
  Myalgia: Post vaccination 2 (Visit 4) | 72 | 70
  Myalgia: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Myalgia: Post CYD vaccination 2 (Visit 5) |  | 43
  Myalgia: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Myalgia: Post CYD vaccination 3 (Visit 7) | 16 | 13
  Asthenia: Post any vaccination: number analyzed (Participants) | 260 | 258
  Asthenia: Post any vaccination | 133 | 132
  Asthenia: Post vaccination 1 (Visit 1): number analyzed (Participants) | 260 | 258
  Asthenia: Post vaccination 1 (Visit 1) | 101 | 89
  Asthenia: Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 255
  Asthenia: Post CYD vaccination 1 (Visit 2) |  | 63
  Asthenia: Post vaccination 2 (Visit 4): number analyzed (Participants) | 256 | 254
  Asthenia: Post vaccination 2 (Visit 4) | 74 | 46
  Asthenia: Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Asthenia: Post CYD vaccination 2 (Visit 5) |  | 35
  Asthenia: Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Asthenia: Post CYD vaccination 3 (Visit 7) | 19 | 16

11. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events Following Vaccination With Gardasil or CYD Dengue Vaccine
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF in terms of diagnosis and/or onset post-vaccination. At Visit 1 and Visit 4, participants from Group 1 received both Gardasil and CYD vaccination and participants from Group 2 received only Gardasil vaccination. At Visit 2 and Visit 5, only participants from Group 2 received CYD vaccination whereas the participants from Group 1 received no vaccination.
Time Frame: Up to 28 days after any and each vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 263 | 260
Participants
  Post any vaccination | 54 | 91
  Post vaccination 1 (Visit 1) | 34 | 38
  Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 256
  Post CYD vaccination 1 (Visit 2) |  | 38
  Post vaccination 2 (Visit 4): number analyzed (Participants) | 257 | 256
  Post vaccination 2 (Visit 4) | 24 | 22
  Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Post CYD vaccination 2 (Visit 5) |  | 28
  Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Post CYD vaccination 3 (Visit 7) | 5 | 7

12. Secondary Outcome: Number of Participants Reporting Non-serious Adverse Event of Special Interests (AESIs) Following Vaccination With Gardasil or CYD Dengue Vaccine
Description: AESI were AEs that were considered by the Sponsor to be relevant for the monitoring of the safety profile of the investigational vaccine. At Visit 1 and Visit 4, participants from Group 1 received both Gardasil and CYD vaccination and participants from Group 2 received only Gardasil vaccination. At Visit 2 and Visit 5, only participants from Group 2 received CYD vaccination whereas the participants from Group 1 received no vaccination.
Time Frame: Within 7 days after any and each vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 263 | 260
Participants
  Post any vaccination | 0 | 0
  Post vaccination 1 (Visit 1) | 0 | 0
  Post CYD vaccination 1 (Visit 2): number analyzed (Participants) | 0 | 256
  Post CYD vaccination 1 (Visit 2) |  | 0
  Post vaccination 2 (Visit 4): number analyzed (Participants) | 257 | 256
  Post vaccination 2 (Visit 4) | 0 | 0
  Post CYD vaccination 2 (Visit 5): number analyzed (Participants) | 0 | 249
  Post CYD vaccination 2 (Visit 5) |  | 0
  Post CYD vaccination 3 (Visit 7): number analyzed (Participants) | 103 | 83
  Post CYD vaccination 3 (Visit 7) | 0 | 0

13. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) Including Serious Adverse Event of Special Interests Following Vaccination With Gardasil or CYD Dengue Vaccine
Description: SAEs were AEs that resulted in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or a medically important event. An AESIs were AEs that were considered by the Sponsor to be relevant for the monitoring of the safety profile of the investigational vaccine.
Time Frame: From Day 0 up to 6 months after the last Gardasil or CYD vaccination
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 263 | 260
Participants
  SAE | 11 | 8
  Serious AESI | 1 | 2

14. Secondary Outcome: Number of Participants Reporting Cases of Virologically Confirmed Dengue (VCD) Hospitalization Following Vaccination With Gardasil or CYD Dengue Vaccine
Description: Hospitalized suspected dengue case was defined as an acute febrile illness with diagnosis of dengue requiring hospitalization (with bed attribution). In such cases, 1 unplanned acute blood sample (within the first 5 days after fever onset) was collected for virological confirmation of hospitalized suspected dengue case. A suspected case was considered VCD if there was a detection of wild type dengue virus by dengue non-structural protein 1 antigen enzyme-linked immunosorbent assay and/or dengue reverse transcriptase-polymerase chain reactions.
Time Frame: From Day 0 up to 6 months after the last Gardasil or CYD vaccination
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
Number analyzed (Participants) | 263 | 260
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: The AE data were collected from Day 0 up to Day 28 post any vaccination. SR were collected from Day 0 up to Day 14 post any vaccination. The SAEs were collected throughout the trial, i.e. 6 months after last Gardasil or CYD vaccination.
Description: The SR was an AE that was prelisted (i.e., solicited) in the electronic CRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF (i.e., solicited) in terms of diagnosis and/or onset post-vaccination. Analysis was performed on SafAS.
Arm/Group | CYD Dengue Vaccine + Gardasil (Concomitant Administration) | CYD Dengue Vaccine + Gardasil (Sequential Administration)
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/260
Serious Adverse Events (participants affected / at risk) | 11/263 | 8/260
Other Adverse Events (participants affected / at risk) | 233/263 | 235/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine + Gardasil (Concomitant Administration) (N=263) | CYD Dengue Vaccine + Gardasil (Sequential Administration) (N=260)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Chikungunya Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Dengue Fever (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gingival Abscess (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sports Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tendon Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Glomerulonephritis Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine + Gardasil (Concomitant Administration) (N=263) | CYD Dengue Vaccine + Gardasil (Sequential Administration) (N=260)
Asthenia (General disorders) | 133 (194) | 132 (249)
Injection Site Erythema (General disorders) | 45 (99) | 38 (63)
Injection Site Pain (General disorders) | 206 (532) | 193 (452)
Injection Site Swelling (General disorders) | 43 (89) | 31 (48)
Malaise (General disorders) | 111 (159) | 137 (260)
Pyrexia (General disorders) | 39 (43) | 53 (61) — Pyrexia events that occurred after 14 days post-vaccination were considered as unsolicited AE.
Upper Respiratory Tract Infection (Infections and infestations) | 20 (21) | 30 (37)
Myalgia (Musculoskeletal and connective tissue disorders) | 127 (181) | 156 (283)
Headache (Nervous system disorders) | 126 (178) | 147 (311) — Headache events that occurred after 14 days post-vaccination were considered as unsolicited AE.

LIMITATIONS AND CAVEATS:
Change of population for non-inferiority reduced to dengue immune participants & time window for 3rd vaccination not reached(study hold),hence non-inferiority analysis not performed & immunogenicity was performed on FAS & not on Per Protocol Set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT02993757/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT02993757/SAP_001.pdf